CLINICAL TRIAL: NCT03436654
Title: Multi-arm Multi-modality Therapy for Very High Risk Localized and Low Volume Metastatic Prostatic Adenocarcinoma
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Dana-Farber Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 17-646; PCCTC #: c16-183 (Other: Prostate Cancer Clinical Trials Consortium, LLC (PCCTC))
Record Dates: First submitted 2018-02-07; First posted 2018-02-19 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Prostate Cancer
Keywords: prostate cancer; apalutamide; abiraterone acetate; memorial sloan kettering cancer center; 17-646
MeSH Terms: conditions — Prostatic Neoplasms | interventions — apalutamide; Abiraterone Acetate; Prednisone; Gonadotropin-Releasing Hormone; Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- ADT + Apalutamide (Experimental)
  Interventions: Drug: Apalutamide; Procedure: Radical Prostatectomy; Procedure: Extended Pelvic lymphadenectomy; Drug: GnRH agonist/antagonist
- ADT + Apalutamide + Abiraterone Acetate + Prednisone (Experimental): This arm is no longer being assigned to subjects.
  Interventions: Drug: Apalutamide; Drug: Abiraterone Acetate; Drug: Prednisone; Procedure: Radical Prostatectomy; Procedure: Extended Pelvic lymphadenectomy; Drug: GnRH agonist/antagonist
- Apalutamide, SBRT, Radiation (Experimental)
  Interventions: Drug: Apalutamide; Radiation: Stereotactic Body Radiation Therapy

INTERVENTIONS:
Drug: Apalutamide — 240mg daily orally
  Other Names: ARN-509, ERLEADA™
Drug: Abiraterone Acetate — 1000mg daily orally
  Other Names: ZYTIGA
  Arms: ADT + Apalutamide + Abiraterone Acetate + Prednisone
Drug: Prednisone — 5mg BID orally
  Arms: ADT + Apalutamide + Abiraterone Acetate + Prednisone
Procedure: Radical Prostatectomy — A laparoscopic, robotic-assisted, or open approach to RP is permitted at the discretion of the operating surgeon.
  Arms: ADT + Apalutamide; ADT + Apalutamide + Abiraterone Acetate + Prednisone
Procedure: Extended Pelvic lymphadenectomy — To be performed concurrently with prostatectomy. Bilateral pelvic lymphadenectomy should include complete removal of all pelvic lymph nodes within the broad template described and includes the external iliac, hypogastric, obturator, and pre-sacral lymph nodes
  Arms: ADT + Apalutamide; ADT + Apalutamide + Abiraterone Acetate + Prednisone
Drug: GnRH agonist/antagonist — Physician's choice, for a total duration not to extend beyond the treatment phase of the protocol or 10 months from the start of investigational agent(s)
  Arms: ADT + Apalutamide; ADT + Apalutamide + Abiraterone Acetate + Prednisone
Radiation: Stereotactic Body Radiation Therapy — Subjects undergo SBRT in cycle 4, then salvage radiation therapy in cycles 7-8. Treatment repeats every 28 days for up to 10 cycles in the absence of disease progression or unacceptable toxicity
  Arms: Apalutamide, SBRT, Radiation

SUMMARY:
The purpose of this study is to test if treatment with medications that reduce the male hormone level in the participant's body for a few months before surgery can shrink prostate cancer as much as possible, which might reduce the chances of the cancer coming back in the future. These treatments include a hormone injection given monthly or every three months and the study drugs, which include abiraterone acetate, prednisone, and apalutamide.

These medications are being used in combination with surgery and maybe radiotherapy because studies have shown that any single approach on its own is not sufficient to control or get rid of the cancer especially if they have high risk or aggressive features. The researchers hope to learn if combining the study drugs with surgery and radiation will get rid of the cancer from participants' prostates and reduce their prostate-specific antigen (PSA) to an undetectable level.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to provide written informed consent and Authorization for Use and Release of Health and Research Study Information (HIPAA authorization) NOTE: HIPAA authorization may be either included in the informed consent or obtained separately
* Male aged 18 years and above
* Serum testosterone of ≥150 ng/dL (For Cohorts A and B1, testosterone level requirement is exempted if they are already on ADT prior to treatment start. For Cohort B2, subjects will be considered eligible if their testosterone is currently ≥150 ng/dl).
* Histologically confirmed adenocarcinoma of the prostate, who meet the following criteria:

Cohort A

* Clinically localized disease with histologically confirmed adenocarcinoma of the prostate with either ≥3 positive cores or 2 positive cores if >1cm in length with at least 50% tumor content WITH
* With Gleason score 8-10 OR
* Gleason 4+3 with one of the following features:
* PSA ≥ 20 mg/mL within 2 months prior to diagnostic biopsy
* MRI suspicious for radiographic ≥T3 disease (if urologist deems tumor is resectable at baseline); defined as >75% probability of extracapsular extension or seminal vesicle invasion in the opinion of the reading radiologist.

OR

* Gleason 3+4 or 4+3 and Oncotype DX Genomic Prostate Score of >40
* With or without clinical N1 (size >1.5cm in the short axis) (Gleason score requirement can be omitted if node positive)

OR

Cohort B1

* Newly diagnosed low-volume metastatic disease with either.
* Bone metastases as documented by CT, MRI or radionuclide bone scan amenable to treatment with a maximum of 3 radiation isocenters* These lesions must have a structural correlate on CT or MRI to allow for adequate radiation targeting

  *(note:subjects with PET scans that show osseous metastases that would not be amenable to 3-isocenter radiation treatment are still eligible if conventional imaging shows osseous disease that can be treated with 3 radiation isocenters) And/or
* Retroperitoneal nodes up to the level of the renal hilum with/without pelvic nodal metastasis >1.5cm in the short axis
* NOTE: For Cohort B1, biopsy confirmation of metastases is strongly encouraged if safe and feasible, but not required

OR

Cohort B2 (Cohort B2 expansion)

* Biochemically persistent/recurrent disease (defined as PSA >0.2) after RP ± extended pelvic nodal dissection with metastatic lesions identified on PSMAb PET scans
* PSMA PET evidence of M1a/M1b disease that could be covered in up to 3 radiation plans (note that the isocenter for planned prostate bed/pelvic nodal irradiation does not count towards the 3 isocenter limit)
* No radiographic evidence of local or regional recurrence on imaging in subjects with prior salvage radiation to these areas.
* Prior salvage radiotherapy is permitted. Prior metastasis-directed radiation is not permitted.
* Castration sensitive disease
* Multiple lesions within one isocenter may be permitted upon review by the sponsor's radiation oncologist
* ECOG performance status of ≤ 1
* NOTE: For Cohort B2, biopsy confirmation of metastases is strongly encouraged if safe and feasible, but not required
* Adequate bone marrow, hepatic and renal function, as evidenced within 28 days prior to treatment start by:

  * ANC ≥ 1500/µl
  * Hemoglobin ≥ 9g/dL
  * Platelet count ≥ 100,000/µl
  * Serum Creatinine GFR ≥30 mL/min
  * Porassium within institutional normal range
  * Total Bilirubin ≤ 1.5 x ULN (Note: In subjects with Gilbert's syndrome, if total bilirubin is >1.5 x ULN, measure direct and indirect bilirubin and if direct bilirubin is ≤ 1.5 x ULN, subject may be eligible)
  * Albumin ≥ 3.0 g/dL
  * SGOT (AST) ≤ 2.5 x ULN
  * SGPT (ALT) ≤ 2.5 x ULN
* Subjects must have a clinical T stage documented by the treating urologist/medical oncologist within 90 days prior to treatment start using the 7th edition AJCC staging system, recorded as the urologist's/medical oncologist's best clinical assessment of extent of local disease by digital rectal examination and/or available imaging studies such as transrectral ultrasound, CT scan, and/or MRI. Applicable to Cohorts A and B1 only.
* The primary tumor must be considered unresectable by RP based on initial imaging with gross negative margins as determined by a urologist and documented as such. (Applicable to Cohorts A and B1 only)
* Recovery of reversible effects of prior surgery (i.e., incisional pain, wound drainage) to Grade ≤1, and at least 4 weeks from prior surgery to treatment start. (biopsy excluded)
* Able to swallow the study drug(s) whole as a tablet
* Willing to take abiraterone acetate on an empty stomach; no food should be consumed at least one hour before and for at least two hours after the dose of abiraterone acetate is taken (Not applicable to Cohort B2 expansion) (Note: apalutamide does not have to be taken on an empty stomach.)
* Agrees to use a condom (even men with vasectomies) and another effective method of birth control if he is having sex with a woman of childbearing potential or agrees to use a condom if he is having sex with a woman who is pregnant while on study drug and for 3 months following the last dose of study drug. Must also agree not to donate sperm during the study and for 3 months after receiving the last dose of study drug.

Exclusion Criteria:

* Prior treatment for prostate cancer including prior surgery (excluding TURP and subjects with rising PSA after RP), pelvic lymph node dissection, and/or radiation therapy unless the subject is eligible for Cohort B2. (Applicable to cohorts A and B1 only).
* Prior cytotoxic chemotherapy or biologic therapy for prostate cancer
* Up to 2 months of prior ADT with GnRH antagonist/agonist at time of treatment start. Bicalutamide given for ≤ 12 months at the time of registration as flare prevention is allowed. For Cohort B2, prior ADT and/or first generation anti-androgen treatment in the (neo)adjuvant and/or salvage setting in conjunction with radiation or surgery is allowed provided last effective dose of ADT and/or first generation anti-androgen is > 12 months prior to the on treatment date and total duration of prior therapy is 12 months or lesser, and their testosterone is currently >150ng/dL.
* Prior exposure to ketoconazole (systemic), abiraterone acetate, enzalutamide or other agents targeting the AR signaling pathway
* Concomitant therapy with any other experimental drug
* Known brain, liver, lung or other visceral metastasis (except for retroperitoneal and/or pelvic nodal metastases as per inclusion criteria)
* Prior prostate cancer metastasis-directed therapies
* Currently active second malignancy or past history of malignancies diagnosed within the last 2 years that require active therapy and/or in remission with life expectancy of < 5 years, with the exception of resected non-melanoma skin cancers, non-muscle invasive bladder cancer, state I head and neck cancer, or stage I colorectal cancer
* Significant medical condition other than cancer, that would prevent consistent and compliant participation in the study that would, in the opinion of the investigator, make this protocol unreasonably hazardous including but not limited to:

  * Any medical condition requiring a higher dose of corticosteroid than 10mg prednisone/prednisolone once daily
  * Active infection requiring systemic therapy
  * History of gastrointestinal disordered (medical disorders or extensive surgery) that may interfere with the absorption of the study agents
  * Uncontrolled hypertension (systolic BP ≥ 160 mmHg or diastolic BP ≥ 95 mmHg); subjects with a history of hypertension are allowed provided blood pressure is controlled by anti-hypertensive treatment (systolic BP < 160 mmHg or diastolic BP <95 mmHg)
  * Active or symptomatic viral hepatitis of chronic liver disease
  * Acute or chronic hepatitis B or hepatitis C infection. (Hepatitis B and C testing are not mandatory)
  * Presence of hepatitis B surface antibody is acceptable

Human immunodeficiency virus (HIV)-positive subjects with 1 or more of the following:

Not receiving highly active anti-retroviral therapy. A change in anti-retroviral therapy within 6 months of the start of screening (except if, after consultation with the principal investigator (PI) / sponsor, a change is made to avoid a potential drug-drug interaction with the study drug).

Receiving anti-retroviral therapy that may interfere with the study drug(s) (consult the PI / sponsor for review of medication prior to enrollment).

CD4 count < 350 cell/mm^3 at screening. An acquired immunodeficiency syndrome-defining opportunistic infection within 6 months of the start of screening.

* History of pituitary or adrenal dysfunction
* History of hypogonadism
* Clinically significant heart disease as evidenced by myocardial infarction, or arterial thrombotic events in the past 6 months, severe or unstable angina, or New York Heart Association (NYHA) Class III or IV heart disease or cardiac ejection fraction measurement of <50% at baseline, or clinically significant ventricular arrhythmias within 6 months prior to treatment start.
* History of seizure or any condition that may predispose to seizure (including, but not limited to prior stroke, transient ischemic attack or loss of consciousness </= 1 year prior to treatment start; brain arteriovenous malformation; or intracranial masses such as schawnnomas and meningiomas that are causing edema or mass effect)
* Uncontrolled diabetes mellitus
* History of inflammatory bowel disease
* Baseline moderate and severe hepatic impairment (Child Pugh Class B & C)

  * Use of any prohibited concomitant medications within 14 days prior to treatment start, or use of prohibited concomitant medication listed in section 7.9.1 within the outlined windows NOTE: Medications known to lower the seizure threshold must be discontinued or substituted at least 4 weeks prior to treatment start
  * Pre-existing condition that warrants long-term corticosteroid use in excess of 10 mg prednisone/prednisolone daily
  * Known allergies, hypersensitivity or intolerance to apalutamide, abiraterone acetate, prednisone, or GnRH agonist or GnRH antagonist (Allergies or hypersensitivity to abiraterone and/or prednisone would not be applicable to subjects enrolling to B2 expansion).
  * Administration of an investigational therapeutic within 30 days of treatment start
  * Patients that cannot tolerate MRI
  * Any condition which, in the opinion of the investigator, would preclude participation in this trial

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Prostate
Enrollment: 102 (Actual)
Dates: Start 2018-06-21 (Actual); Primary Completion 2026-02-14 (Estimated); Study Completion 2026-02-14 (Estimated)

PRIMARY OUTCOMES:
Pathologic complete response | 24 months
  The primary efficacy measure of pathological complete response and minimal residual disease is defined as the less than or equal to 5 mm of morphologically identifiable carcinoma in the RP specimen.
Minimal residual disease (MRD) | 24 months
  ≤ 5mm tumor

SECONDARY OUTCOMES:
PSA Response Rate | 10 months from randomization
  defined as percentage of patients with an undetectable PSA at 10 months from randomization (after completion of all protocol treatment)
Time to PSA Progression | 24 months
  Time from the start of treatment to the date of first evidence of disease progression (serum PSA ≥0.2ng/mL, which is confirmed by a second determination with a PSA ≥0.2 ng/mL, according to the 2007 American Urological Association Prostate Guidelines). This will be estimated by the cumulative incidence function. For each arm, time to PSA progression will be presented for all patients as well as by metastatic status

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Dallos, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (11):
- United States (11):
  - University of Chicago, Chicago, Illinois
  - Northwestern University, Evanston, Illinois
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Memorial Sloan Kettering Basking Ridge (Limited Protocol Activities), Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth (Limited Protocol Activities), Middletown, New Jersey
  - Memorial Sloan Kettering Bergen (Limited Protocol Activities), Montvale, New Jersey
  - Memorial Sloan Kettering Commack (Limited Protocol Activities), Commack, New York
  - Memorial Sloan Kettering Westchester (Limited Protocol Activities), Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering Nassau (Limited Protocol Activities), Uniondale, New York
  - Cleveland Clinic, Cleveland, Ohio

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://mskcc.org